CLINICAL TRIAL: NCT02721537
Title: Use of 31P MRS to Assess Brain NAD+ in Healthy Current and Former Collegiate Athletes and a Comparison of the Effect of Nicotinamide Riboside Supplementation on Brain NAD+ Levels
Brief Title: Use of 31P MRS to Assess Brain NAD+ in Healthy Current and Former Collegiate Athletes
Acronym: TRMC-004
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: University of Minnesota (Other); Thorne HealthTech, Inc (Industry)
Responsible Party: Principal Investigator, Brent A. Bauer, M.D., Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 15-006870
Record Dates: First submitted 2016-03-24; First posted 2016-03-29 (Estimated); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Concussion, Mild
Keywords: Brain Nicotinamide Adenine Dinucleotide (NAD+); Adenosine Triphosphate (ATP) Depletion; Polyadenosine Diphosphate-Ribosepolymerase (PARP) Activation
MeSH Terms: conditions — Brain Concussion | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: Healthy Collegiate Athletes (Active Comparator): Healthy collegiate athletes will take active Nicotinamide Riboside
  Interventions: Dietary Supplement: Nicotinamide Riboside
- Arm B: Healthy Collegiate Athletes (Placebo Comparator): Healthy collegiate athletes will take a matching placebo
  Interventions: Other: Matching placebo

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside — Three capsules, twice per day for 84 days
  Other Names: Niagen
  Arms: Arm A: Healthy Collegiate Athletes
Other: Matching placebo — Three matching capsules, twice per day for 84 days
  Arms: Arm B: Healthy Collegiate Athletes

SUMMARY:
Can nicotinamide riboside (750 mg/day for 12 weeks) affect the levels of NAD+ in the brain as measured by 31P MRS?

DETAILED DESCRIPTION:
Healthy collegiate athletes (football, soccer, rugby, hockey, and volleyball) will take Nicotinamide Riboside (NR) or placebo twice daily for 84 days. Pre- and post-intervention evaluations include physical assessment, blood tests for safety and toxicity monitoring, blood tests for biomarkers, neurologic testing, quality of life questionnaires, and the 31P MRI exam.

ELIGIBILITY:
Inclusion Criteria:

* Adult current and former (within 2 years) collegiate athletes (football, rugby, soccer, hockey, and volleyball)
* Body mass index (estimated based on height and weight) from 23 to 37
* Willing to provide informed consent, ingest test substance, and provide blood specimens
* Willing to comply with study instructions and maintain current level of physical activity throughout the study

Exclusion Criteria:

* History of loss of consciousness of more than 5 minutes
* Contraindications to Magnetic Resonance Imaging (MRI), such as implanted medical devices, metal objects, or pacemakers
* History of epilepsy
* History of more than 3 concussions
* History of headache preceding a concussion
* History of depression preceding a concussion
* History of developmental delays or Attention Deficit Hyperactivity Disorder (ADHD)
* History of post-traumatic seizures
* History of complex spine and/or skull trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-09; Primary Completion 2022-08 (Actual); Study Completion 2022-08 (Actual)

PRIMARY OUTCOMES:
Change in brain NAD+ levels | baseline, day 84
  As measured by 31P MRI

CONTACTS AND LOCATIONS:
Overall Officials: Brent A Bauer, MD, Principal Investigator — Mayo Clinic in Rochester, MN
Locations (2):
- United States (2):
  - University of Minnesota Center for Magnetic Resonance Research, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials